CLINICAL TRIAL: NCT05340465
Title: Trial of Darbepoetin Plus Slow-release Intravenous Iron to Decrease Transfusions and Improve Iron Status and Neurodevelopment in Preterm Infants
Brief Title: Darbe Plus IV Iron to Decrease Transfusions While Maintaining Iron Sufficiency in Preterm Infants
Acronym: DIVI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kendell German, Associate Professor: School of Medicine, Pediatrics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00015143; R01HD107003 (NIH)
Record Dates: First submitted 2022-03-01; First posted 2022-04-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prematurity; Iron-deficiency; Iron Deficiency Anemia; Iron Malabsorption
Keywords: prematurity; iron deficiency; anemia; darbepoetin; IV Iron
MeSH Terms: conditions — Premature Birth; Anemia, Iron-Deficiency; Iron Deficiencies; Anemia | interventions — Darbepoetin alfa; Iron-Dextran Complex; Ferrosoferric Oxide

STUDY DESIGN:
Intervention Model Description: * Group 1 Control, oral iron up to 12 mg/kg/day per Unit protocol
  * Group 2 Darbe 10 mcg/kg q week plus LMW-ID: 10 mg/kg x 1, retreat if ferritin < 76 mcg/L
  * Group 3 Darbe 10 mcg/kg q week plus LMW-ID: 20 mg/kg x 1, retreat if ferritin < 76 mcg/L
  * Group 4 Darbe 10 mcg/kg q week plus FMX 10 mg/kg x 1, retreat if ferritin < 76 mcg/L
  * Group 5 Darbe 10 mcg/kg q week plus FMX 20 mg/kg x 1, retreat if ferritin < 76 mcg/L
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Group 1 will be unblinded. In Groups 2-5 all infants will receive Darbe, and the iron preparation and dose will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 1. Oral iron (Active Comparator): Oral iron is started on day 7 of life if baby is feeding 100 mL/kg/day. Iron supplements of up to 12 mg/kg/day are given based on CBC, retic, ret-hgb, serum ferritin and zinc protoporphyrin to heme ratio (ZnPP/H). Iron supplements are adjusted every 2 weeks following iron studies.
  Interventions: Drug: Oral iron supplements
- Group 2 (Experimental): Infants randomized to this arm will receive Darbe 10 mcg/kg q week started on day 3 of life. In addition, beginning on day 7, they will receive LMW-ID: 10 mg/kg x 1, retreat if ferritin < 76 mcg/L
  Interventions: Drug: Darbepoetin Alfa; Drug: Low Molecular Weight Iron Dextran
- Group 3 (Experimental): Infants randomized to this arm will receive Darbe 10 mcg/kg q week started on day 3 of life. In addition, beginning on day 7, they will receive LMW-ID: 20 mg/kg x 1, retreat if ferritin < 76 mcg/L
  Interventions: Drug: Darbepoetin Alfa; Drug: Low Molecular Weight Iron Dextran
- Group 4 (Experimental): Infants randomized to this arm will receive Darbe 10 mcg/kg q week started on day 3 of life. In addition, beginning on day 7, they will receive FMX: 10 mg/kg x 1, retreat if ferritin < 76 mcg/L
  Interventions: Drug: Darbepoetin Alfa; Drug: Ferumoxytol injection
- Group 5 (Experimental): Infants randomized to this arm will receive Darbe 10 mcg/kg q week started on day 3 of life. In addition, beginning on day 7, they will receive FMX: 20 mg/kg x 1, retreat if ferritin < 76 mcg/L
  Interventions: Drug: Darbepoetin Alfa; Drug: Ferumoxytol injection

INTERVENTIONS:
Drug: Darbepoetin Alfa — Infants in groups 2-5 will be started on Darbe 10 mcg/kg/week between 72 and 84 hours after birth.
  Other Names: Aranesp; Darbe
  Arms: Group 2; Group 3; Group 4; Group 5
Drug: Low Molecular Weight Iron Dextran — Infants in groups 2 and 3 will be given LMW-ID IV, 10 or 20 mg/kg/dose. They will be re-dosed if ferritin falls below 76. Iron parameters will be checked biweekly.
  Other Names: INFeD; LMW-ID
  Arms: Group 2; Group 3
Drug: Ferumoxytol injection — Infants in groups 4 and 5 will be given FMX IV, 10 or 20 mg/kg/dose. They will be re-dosed if ferritin falls below 76. Iron parameters will be checked biweekly.
  Other Names: Feraheme; FMX
  Arms: Group 4; Group 5
Drug: Oral iron supplements — Infants in group 1 will receive standard care in the UW NICU with iron started on day 7 if tolerating 100 mL/kg/day enteral feeding. Iron supplements are adjusted every 2 weeks based on ferritin, zinc protoporphyrin to heme ratio and complete blood count (CBC).
  Other Names: Ferr-in-sol
  Arms: Group 1. Oral iron

SUMMARY:
In this phase II trial, the investigators overarching goal is to demonstrate the feasibility and potential benefit of darbepoetin (Darbe) plus slow-release intravenous (IV) iron to decrease transfusions, maintain iron sufficiency and improve the neurodevelopmental outcomes of preterm infants.

Investigators hypothesize that in infants < 32 completed weeks of gestation, combined treatment with Darbe plus Ferumoxytol (FMX) or Darbe plus low molecular weight iron dextran (LMW-ID) will: 1) be safe, 2) decrease or eliminate transfusions, 3) maintain iron sufficiency, 4) result in higher hematocrit and 5) improve neurodevelopment. Investigators further hypothesize that when compared to oral iron supplementation (standard care), IV iron will be better tolerated, with less effect on the gastrointestinal (GI) microbiome

DETAILED DESCRIPTION:
Investigators hypothesize that in infants < 32 completed weeks of gestation, combined treatment with Darbe plus FMX or Darbe plus LMW-ID will: 1) be safe, 2) decrease or eliminate transfusions, 3) maintain iron sufficiency, 4) result in higher hematocrit and 5) improve neurodevelopment. Investigators further hypothesize that when compared to oral iron supplementation (standard care), IV iron will be better tolerated, with less effect on the gastrointestinal (GI) microbiome

Objectives:

1. To compare the safety, dose, and dosing interval for FMX and LMW-ID required for preterm infants receiving Darbe.

   Iron dosing will begin at 7 days after birth. Initial doses of 10 mg/kg/dose or 20 mg/kg/dose will be compared for each iron formulation (N=20 each).
2. To compare the safety, tolerance, and efficacy of IV iron (FMX or LMW-ID) plus Darbe (N=80) to standard care (oral ferrous sulfate (N=40). Adverse reactions to IV Iron will be documented, as will adverse responses to oral iron (feeding intolerance). Potential differences in the stool microbiome will be evaluated 3 weeks after the initial IV and oral iron doses.
3. Determine long-term outcomes:

   * 3.1 Neurodevelopmental outcomes of infants enrolled in Objectives 1 and 2 (N=120) will be sequentially assessed up to 2 years of age.
   * 3.2 The stool microbiome will be compared between study groups at 12 and 24 months to determine whether mode of iron delivery has long-term effects.

ELIGIBILITY:
Inclusion Criteria:

• NICU patients (male and female) born at 24-0/7 to 31-6/7 weeks of gestation

All patients who meet inclusion criteria will be approached without regard to sex, race, ethnicity, parents' country of origin, or religious preferences.

Exclusion Criteria:

* Known fetal/infant anomalies of clinical significance (brain, cardiac, chromosomal anomalies)
* Parental consent unable to be obtained by 72 hours after birth
* Central hematocrit > 65%
* Evidence of high iron stores prior to enrollment (e.g. Ferritin >400 ng/mL with corresponding ZnPP/H of <30, Transferrin saturation >75%, iron > 200 mcg/dL, TIBC < 100 mcg/dL)
* Culture proven sepsis, meningitis, urinary tract infection, or other significant infection at the time of enrollment
* Mother under 18 years of age
* Unable to consent in English or Spanish

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-11-27 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Plasma Ferritin at 35-36 weeks PMA | birth to 36 weeks postmenstrual age
  Plasma ferritin is measured every 2 weeks in the NICU. Ferritin at 35-36 weeks will be compared between the 5 treatment groups
Number of IV iron doses required to maintain a ferritin level of > 75 ng/mL | Birth to 36 weeks postmenstrual age (or prior to discharge if this occurs prior to 36 weeks)
  Number of IV iron doses required to maintain a ferritin level of > 75 ng/mL will be compared in the 4 IV treatment arms
Number of Blood transfusions | Birth to 36 weeks postmenstrual age (or prior to discharge if this occurs prior to 36 weeks)
  The number of blood transfusions received by infants in each group will be compared.
Volume of blood transfusions | Birth to 36 weeks postmenstrual age (or prior to discharge if this occurs prior to 36 weeks)
  The volume of blood transfused to infants in each group will be compared

SECONDARY OUTCOMES:
Number and percent of patients per group that remain transfusion free | Birth to 36 weeks postmenstrual age (or prior to discharge if this occurs prior to 36 weeks)
  Number and percent of patients per group that remain transfusion free will be compared by group
Hematocrit | Birth to 36 weeks PMA
  Hematocrit (lowest, highest, mean) by group to 35-36 weeks PMA
Safety of IV iron | Birth to 36 weeks postmenstrual age (or prior to discharge if this occurs prior to 36 weeks)
  Any evidence of anaphylaxis will be documented during and after the first IV infusion of iron
Early gut microbiome comparison between study groups | at 7 days (prior to iron supplementation) and 4 weeks after birth
  Stool samples will be collected for 16S amplicon sequencing and targeted culturomics. Organism types will be compared between groups prior to and 3 weeks after the first IV iron dose.
Rate of referral for Brainstem auditory evoked response | at hospital discharge, near 36 weeks postmenstrual age
  Any latency in Brainstem auditory evoked response will be assessed and compared between study arms
Rate of pass/fail the General Movements Assessments (GMA) | 3 months corrected age
  General Movements Assessments (GMA) will be assessed at 3 months corrected age, and results compared between study arms.
Scores for the Warner Initial Developmental Evaluation of Adaptive and Functional Skills (WIDEA-FS) will be compared between groups | 6 months corrected age
  Parent questionnaire (WIDEA-FS) to assess neurodevelopment will be done at 6 months corrected age. Mean and median scores will be compared by treatment arm. The WIDEA includes 50 items with a maximum score of 200. Higher scores indicate more advanced neurodevelopmental functioning.
Scores for the Warner Initial Developmental Evaluation of Adaptive and Functional Skills (WIDEA-FS) will be compared between groups | 18 months corrected age
  Parent questionnaire (WIDEA-FS) to assess neurodevelopment will be done at 6 months corrected age. Mean and median scores will be compared by treatment arm. The WIDEA includes 50 items with a maximum score of 200. Higher scores indicate more advanced neurodevelopmental functioning.
Late gut microbiome comparison between study groups | at 1 and 2 years corrected age.
  Stool samples will be collected for 16S amplicon sequencing and targeted culturomics. Organism types will be compared between groups. If differences in early microbiome (at 4 weeks of age) are noted, we will evaluate whether they persist at 1 and 2 years of age.
Neurodevelopmental outcome as assessed by the Bayley Scales of Infant Development edition-IV (BSID-IV) | 1 year and 2 years corrected age
  Bayley Scales of Infant Development edition-IV (BSID-IV) will be assessed in all enrolled patients at one and two years corrected age. Results for the treatment arms will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Kendell R German, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We will comply with and share data in accordance with the definitions contained in the guidance document:
  Data Element Definitions for Interventional and Observational Studies (https://prsinfo.clinicaltrials.gov/results_definitions.html) and the final rule (42 CFR Part 11) .
  In addition, we will comply with NICHD requirements to release our de-identified data-set to the Data and Specimen Hub (DASH), a centralized resource for researchers to store and access data from studies funded by NICHD after the acceptance of publication of our main findings of the final data set (2 year outcomes) as per the NIH Data Sharing Policy: https://dash.nichd.nih.gov/. Biospecimens will not be available. Data will include study protocol, CRFs, and collected, de-identified data collected in REDCap.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 12 months of publication of our primary outcome, a final study data set will be accessible via a supervised private data enclave. Access will be limited to registered users who submit proposed specific questions or analysis plans and sign a data use agreement. "Supervised" indicates that individual requests are reviewed to protect the intellectual property rights of the project investigative team by restricting external development of manuscripts using the study data that substantially overlap with those that are already in development by study investigators. We will form a publications committee, with investigator representatives from the Clinical Coordinating Center and Data Coordinating Center at the University of Washington to establish manuscript development and publication guidelines.
Access Criteria: We will electronically document data requests through a web-based data portal at the University of Washington Center for Biomedical Statistics. The final research data set will be stored separately from the operational study database in a secure web-accessible REDCap database (at https://rcnut.iths.org), where access and downloads can be easily monitored and the data are downloadable in a variety of formats (Excel, R, SAS, Stata, SPSS). A comprehensive data dictionary will be available alongside the final research database. The data sharing plan will be executed within the final year of funding. The overhead required to support this data sharing plan is minimal and therefore no additional budget is requested to cover its costs.

REFERENCES:
- [Derived] Juul SE, Comstock BA, Mayock DE, German K, Feltner J, Irvine J, Lagerquist E, Heagerty PJ. Darbepoetin plus slow-release IntraVenous Iron to decrease transfusions and improve iron status and neurodevelopment in preterm infants (DIVI): study protocol for a randomized, blinded phase II trial. Trials. 2025 Dec 22;26(1):590. doi: 10.1186/s13063-025-09374-9. PMID 41430711